CLINICAL TRIAL: NCT01803802
Title: Effects of Early Abuse on Adult Intimate Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tierney Kyle Ahrold Lorenz, Study Coordinator, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01HD051676 (NIH); R01HD051676 (NIH)
Record Dates: First submitted 2013-02-25; First posted 2013-03-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Hypoactive Sexual Desire Disorder; Female Sexual Arousal Disorder; Female Orgasmic Disorder; Major Depressive Disorder; Post-traumatic Stress Disorder
Keywords: childhood sexual abuse; depression; PTSD; sexual function; women
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Time management (Placebo Comparator): Writing prompts oriented towards objective recounting of previous day
  Interventions: Behavioral: Expressive writing
- Sexual schema writing (Experimental): Expressive writing prompts oriented towards beliefs about sexuality
  Interventions: Behavioral: Expressive writing
- Trauma writing (Active Comparator): Expressive writing prompts oriented towards processing traumatic experiences
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — Five sessions of 30 minutes of expressive writing

SUMMARY:
This study is designed to help us better understand the factors that affect the sexual lives of women who have been sexually mistreated during childhood. With this study we hope to learn about factors that may be promising targets for future treatments of sexual problems related to past sexual experiences. The investigators hypothesize that women who have experienced early sexual abuse are more likely to have sexual problems in adulthood than women who were not abuse in childhood.

ELIGIBILITY:
Inclusion Criteria:

* at least one involuntary sexual experience, defined as "unwanted oral, anal, or vaginal intercourse, penetration of the vagina or anus using objects or digits, or genital touching or fondling," before age 16 and no less than 2 years prior to enrollment.
* currently sexually active or cohabiting in a potentially sexual relationship.
* current sexual dysfunction, distress, or low sexual satisfaction

Exclusion Criteria:

* traumatic event in the previous three months
* sexual abuse in the past two years
* diagnosis of a psychotic disorder in the previous six months
* significant suicidal or homicidal intent
* currently receiving psychotherapy for sexual or abuse-related concerns
* use of illicit drugs
* in a currently abusive relationship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-04; Primary Completion 2011-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sexual Dysfunction Interview | 6 months
  Clinical classification of Female Sexual Dysfunctions including Hypoactive Sexual Desire Disorder, Female Sexual Arousal Disorder, and/or Female Orgasm Disorder

SECONDARY OUTCOMES:
Depression | 6 months
  As measured by clinical interview and validated questionnaires
Post-Traumatic Stress | 6 months
  As measured by clinical interview and validated questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Meston CM, Lorenz TA, Stephenson KR. Effects of expressive writing on sexual dysfunction, depression, and PTSD in women with a history of childhood sexual abuse: results from a randomized clinical trial. J Sex Med. 2013 Sep;10(9):2177-89. doi: 10.1111/jsm.12247. Epub 2013 Jul 22. PMID 23875721
- See also: Link to laboratory website — http://mestonlab.com